CLINICAL TRIAL: NCT04901936
Title: An Open Label, Single-Arm, Phase 2 Study to Evaluate the Safety, Pharmacokinetics, and Biologic Activity of Pegcetacoplan in Pediatric Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: A Study of Pegcetacoplan in Pediatric Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL2-PNH-209
Record Dates: First submitted 2021-03-08; First posted 2021-05-26 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH); Paroxysmal Hemoglobinuria
Keywords: Paroxysmal Nocturnal Hemoglobinuria; PNH; Pediatric; Adolescent; Apellis; Anemia, Hemolytic; Pegcetacoplan; APL-2
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Anemia, Hemolytic | interventions — pegcetacoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pegcetacoplan (Experimental)
  Interventions: Drug: Pegcetacoplan

INTERVENTIONS:
Drug: Pegcetacoplan — Complement (C3) inhibitor

SUMMARY:
The purpose of this study is to evaluate the safety, effectiveness, and biological activity (how the investigational medication is processed by the body) of pegcetacoplan in 12-17 year-olds (adolescents) who have paroxysmal nocturnal hemoglobinuria (PNH).

DETAILED DESCRIPTION:
This is an open-label study to evaluate pegcetacoplan in people with PNH who are 12-17 years old. The study will consist of a 4-week screening period followed by a 16-week treatment period. Participants switching from a C5 inhibitor will have an additional 4 week run-in period between the screening and treatment periods. At the completion of the study treatment period, participants will either enter a long-term extension period or a 2-month follow-up period.

All eligible study participants will receive pegcetacoplan, administered via subcutaneous infusion twice a week at home. The subcutaneous infusion requires two small needles to be inserted into the fatty layer of tissue under the skin and the investigational medication will flow into the body. Study participants and/or caregivers will be trained on home administration of pegcetacoplan.

ELIGIBILITY:
Inclusion Criteria:

* Are 12-17 years old at the time of screening
* Weigh at least 20 kg (approx. 44 lbs)
* Have the diagnosis of PNH, confirmed by high-sensitivity flow cytometry (granulocyte or monocyte clone >10%)
* EITHER:

  * Not being treated with an approved complement inhibitor (eculizumab or ravulizumab) prior to start of pegcetacoplan dosing, AND have hemolytic anemia. Hemolytic anemia is defined as hemoglobin (Hb) less than the lower limit of normal (Hb < LLN) and LDH >1.5 times the upper limit of normal (ULN); OR
  * Currently receiving treatment with an approved complement inhibitor (eculizumab or ravulizumab) AND have evidence of ongoing anemia. Ongoing anemia is defined as Hb < LLN and ARC > ULN
* Have a platelet count >75,000/mm3 and an absolute neutrophil count >1000/mm3

Exclusion Criteria:

* Are an adult, 18 years of age or older, with PNH
* Known or suspected hereditary fructose intolerance (HFI)
* History of hereditary complement deficiency, bone marrow transplant, or meningococcal disease (meningitis, bacteremia or septicemia)
* Females who are pregnant or breastfeeding

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pegcetacoplan serum concentrations over the course of the 16-week treatment period | 16 weeks
Change from baseline to Wk 16 in hemoglobin (Hb) | 16 weeks
Incidence and severity of treatment-emergent adverse events (TEAEs) over the course of the 16-week treatment period, including monitoring bacterial infections | 16 weeks
Change from baseline to wk 16 lactate dehydrogenase (LDH) | 16 weeks
Change from baseline to wk 16 absolute reticulocyte count (ARC) | 16 weeks

SECONDARY OUTCOMES:
Change from baseline from week 16 to week 52 of C3 deposition on RBC cells | Week 16-52
Incidence of thromboembolic events (major adverse vascular events [MAVE]) over the course of the 16-week treatment period and over 52 weeks of treatment with pegcetacoplan | 52 weeks
Occurrence of breakthrough hemolysis over 16 and 52 weeks of treatment with pegcetacoplan | Week 16-52
Change from baseline to Week 52, and from Week 16 to Week 52 , in Hb | Week 16-52
Change from baseline to Week 16 and to Week 52 in Health-Related Quality of Life (HRQOL) assessments | Week 16-52
Number of packed red blood cell (PRBC) units | Week 16-52
Total units (mL/kg) transfused over 16 and 52 weeks of treatment with pegcetacoplan | Week 16-52
Change from baseline to Week 52, and from Week 16 to Week 52, in LDH | Week 16-52
Change from baseline to Week 52, and from Week 16 to Week 52 ARC | Week 16-52

CONTACTS AND LOCATIONS:
Locations (12):
- Children's Hospital of Atlanta, Atlanta, Georgia, United States
- Motol University Hospital, Prague, Czechia
- Robert-Debré Hospital Paris, Paris, France
- Hospital Ampang, Ampang, Malaysia
- Netherlands (2):
  - Radboud University Hospital Nijmegen, Nijmegen
  - University Medical Center Utrecht, Utrecht
- University Children's Hospital, Belgrade, Serbia
- Spain (2):
  - University Hospital Vall d'Hebron, Barcelona
  - University Hospital 12 de Octubre, Madrid
- Thailand (2):
  - Phramongkutklao Hospital and College of Medicine, Bangkok
  - Maharaj Nakorn Chiang Mai hospital, Chiang Mai
- St. Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No